CLINICAL TRIAL: NCT05319223
Title: Patient Blood Management in Orthopedic Surgical Patients in Turkey
Acronym: PABMOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prof. Serdar Gunaydin (Other)
Responsible Party: Sponsor-Investigator, Prof. Serdar Gunaydin, Prof. Dr, ERAS Turkey Association
Organization: ERAS Turkey Association (Other)
Other Study IDs: 110-627-21
Record Dates: First submitted 2022-02-28; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Arthropathy
Keywords: Arthroplasty; patient blood management; anemia; İron deficiency
MeSH Terms: conditions — Joint Diseases; Anemia; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient management group: patient blood management group
  Interventions: Behavioral: patient blood management
- Control: control

INTERVENTIONS:
Behavioral: patient blood management — three pillars of patient blood management will be applied
  Groups: Patient management group

SUMMARY:
Transfusion practice for surgical patients has changed from replacing surgically lost blood with allogeneic blood transfusions to implementing strategies that reduce transfusion requirements. Patient Blood Management (PBM), which is "the timely application of evidence-based medical and surgical concepts designed to maintain haemoglobin concentration, optimize hemostasis and minimize blood loss in an effort to improve patient outcome. There is mounting evidence that multimodal patient blood management (PBM) programmes can be effective at improving postoperative outcomes and reducing perioperative blood transfusions and costs The Turkish Society of Anaesthesiologists PBM Task Force has been working on this subject and studied transfusion practice throughout all through the peri-operative periods. Unfortunately we documented a high transfusion rate in major surgical patients in Turkey. One of the surgeries, that has high transfusion rate, was orthopaedic surgery. According to our recent data we planned to implement PBM in major orthopaedic surgical patients and evaluate the effects PBM in transfusion rate and patient outcomes. While some elements of PBM have a strong evidence base in hip or knee replacement, such as the use of tranexamic acid (TXA) the evidence for preoperative anaemia optimisation with iron is less robust. Implementing PBM all through the operative period gains more importance.

DETAILED DESCRIPTION:
Active PBM Implementation: Patients undergoing hip or knee arthroplasty will be treated as follows: PBM will be performed as shown in the graph below "PBM Implementation Group".

Active PBM group will be treated for preoperative anemia at least 3 weeks prior to the surgical intervention as per the "Anemia Algorithm" below Other pillars of PBM will be also performed to the treatment group as per the visual graph below. The parameters included in the PBM pillars will be recorded including preoperative anemia parameters. Postoperative variables and parameters related to complications will be recorded.

For the control group (Non-PBM group), the data of the patients, will be prospectively included.

The 1:1 ratio of the control and active groups will be done.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this trial, an individual must meet all of the following criteria:

* Signed patient informed consent
* Male or female patient at least 18 years old
* Patients scheduled for an elective major orthopaedic surgery (hip arthroplasty, knee arthroplasty, primary and revision operations)
* Patients with confirmed iron deficiency anemia (IDA), defined as Hb 100-130 g/L, and serum ferritin < 100 ng/ml or TSAT < 20%.

Patients with iron deficiency anemia will be taken into surgery at least 3 weeks after the treatment.

Exclusion Criteria:

* Patients that undergo emergency surgical procedure and trauma cases are excluded from the study.
* Patients with non-iron deficiency anaemia (thalassemia, sickle cell anaemia and etc.)
* Patients with renal anaemia (Hb < 130 g/L and CCL < 50 mL/min, irrespective of iron parameters) or any diagnosis that require EPO will be excluded
* Patients with known anaphylactic/hypersensitivity reactions to parenteral iron products.
* Patients with iron overload or disturbances in utilization of iron (e.g. haemochromatosis, hemosiderosis)
* Patients with ≥3 times increase in aspartate aminotransferase or alanine aminotransferase as per reference range.
* Patients with excessive blood loss requiring massive transfusion (≥ 10 more red blood cell units)
* Patients with known myelodysplastic syndromes.
* Patients with chronic kidney disease with an estimated GFR < 30 ml/min or with end-stage renal disease requiring scheduled dialysis.
* Patients with known urinary tract infections with urea-splitting bacteria
* Any patient judged to lack the ability to give informed consent or perform the trial assessments (e.g. due to dementia)
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases (Female participants who are surgically sterilized / hysterectomized or post-menopausal for longer than 2 years are not considered as being of child bearing potential),
* Known or suspected non-compliance, drug or alcohol abuse,
* Participation in another study with investigational drug within the 30 days preceding and during the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing arthroplasty with anemia
Sampling Method: Non-Probability Sample
Enrollment: 369 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
red cell transfusion | 3 days
  change in red blood cell transfusion rate

SECONDARY OUTCOMES:
cost | 3 days
  change in total hospital cost

CONTACTS AND LOCATIONS:
Overall Officials: Cigdem YILDIRIM GUCLU, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided